CLINICAL TRIAL: NCT00845416
Title: Newborn Screening for SCID in a High-Risk Population
Brief Title: Newborn Screening for Severe Combined Immunodeficiency (SCID) in a High-Risk Population
Status: Completed | Type: Observational
Sponsor: University of California, San Francisco (Other)
Responsible Party: Sponsor
Other Study IDs: H55235-32562-01; R03HD060311 (NIH)
Record Dates: First submitted 2009-02-17; First posted 2009-02-18 (Estimated); Last update posted 2012-07-16 (Estimated); Status verified 2012-07

CONDITIONS: Severe Combined Immunodeficiency; T Cell Lymphocytopenia
Keywords: TREC; T cell; Primary Immunodeficiency; PID; Navajo; SCID
MeSH Terms: conditions — Severe Combined Immunodeficiency; Primary Immunodeficiency Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The goal of the proposed research is to establish the validity of a newborn screening method for severe combined immunodeficiency (SCID). The assay to be used is developed on the basis of PCR quantification of T-cell receptor excision circles (TRECs) that is absent in SCID patients, thus correlating with the disease

DETAILED DESCRIPTION:
To show that early diagnosis of SCID with a TREC screening assay can warrant timely treatment of the disease and avoid life-threatening infections on patients. Babies with SCID are unable to fight infections. They become severely ill in their first months of life and do not survive unless their immune systems can be restored. SCID can be treated by bone marrow transplant if recognized early. The newborn screening test to be employed in this study is designed to diagnose SCID before infections occur. By conducting a pilot testing program in a high-risk population on the Navajo Indian Reservation, where one in 2,000 infants is born with SCID, we hope to confirm the benefits of newborn screening for early diagnosis of SCID

ELIGIBILITY:
Inclusion Criteria:

* Birth in a study hospital on the Navajo Reservation

Exclusion Criteria:

* None

Ages: 1 Day to 30 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Navajo Indians
Sampling Method: Non-Probability Sample
Enrollment: 1800 (Actual)
Dates: Start 2009-03; Primary Completion 2011-11 (Actual); Study Completion 2011-11 (Actual)

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Chinle Hospital, Chinle, Arizona
  - Tuba City Hospital, Tuba City, Arizona